CLINICAL TRIAL: NCT03284086
Title: Comparison of Peak Oxygen Uptake and Exercise Efficiency Between Upper-body Poling and Arm Crank Ergometry in Trained Paraplegic and Able-bodied Participants
Brief Title: VO2peak and Exercise Efficiency in Upper-body Poling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015/2008
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Spinal Cord Injuries
Keywords: Oxygen consumption; Physical endurance
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- paraplegic (Other): Well-trained participants with a spinal cord injury (<Th1) were included in this group.
  Interventions: Diagnostic Test: upper-body double-poling; Diagnostic Test: arm crank ergometry
- able bodied (Other): Upper-body trained, able-bodied participants were included in this group.
  Interventions: Diagnostic Test: upper-body double-poling; Diagnostic Test: arm crank ergometry

INTERVENTIONS:
Diagnostic Test: upper-body double-poling — An incremental peak test to exhaustion and four 5-min submaximal stages were performed in the upper-body double-poling mode.
Diagnostic Test: arm crank ergometry — An incremental peak test to exhaustion and four 5-min submaximal stages were performed in the arm crank ergometry mode.

SUMMARY:
This study compares peak oxygen uptake (VO2peak) and exercise efficiency in upper-body poling versus arm crank ergometry in trained able-bodied and paraplegic participants.

DETAILED DESCRIPTION:
Peak oxygen uptake (VO2peak) and exercise efficiency are key factors for endurance performance. In persons who are primarily able to use their upper-body during exercise, such as many Paralympic athletes, the mode most commonly used in assessing VO2peak and efficiency is arm crank ergometry (ACE). However, sport-specificity of the test mode has been suggested to be of importance for achieving VO2peak and exercise efficiency that are reflective of the aerobic capacity in the respective sport. For ice sledge hockey players, cross-country sit skiers and sitting biathletes, upper-body poling (UP) is the most sport-specific test mode. However, it has not yet been investigated whether VO2peak and efficiency differ between ACE and UP. Therefore, the aim of this study was to compare VO2peak and exercise efficiency in upper-body poling versus arm crank ergometry in trained able-bodied and paraplegic participants. Participants performed four 5-min submaximal stages at increasing effort and an incremental peak test to exhaustion in both ACE and UP.

ELIGIBILITY:
Inclusion Criteria:

* participants between the age of 18 and 50
* well upper-body-trained participants with or without paraplegia

Exclusion Criteria:

* people with injuries or sicknesses that might have impacted the testing

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake | 3 weeks
  Peak oxygen uptake was measured during an incremental test to exhaustion.

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn Helbostad, phd prof, Study Director — Dept of Neuromedicine and Movement Science, Norwegian University of Science and Technology
Locations (1):
- Centre for Elite Sports Research, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes
All data will be de-identified by the project coordinator. The de-identified data will be stored on the NTNU server in a folder that only the JKB and ØS have access to. For analysing the data, parts of the de-identified data might be distributed amongst the four researchers and two master students linked to this study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: September 2016-May 2017